CLINICAL TRIAL: NCT01487278
Title: Preventing Postpartum Hemorrhage: Examining Two Strategies for PPH Prevention in Communities: Misoprostol and Oxytocin in UnijectTM in Mali
Brief Title: Comparing Misoprostol and Oxytocin in UnijectTM for Postpartum Hemorrhage (PPH) Prevention in Mali
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: The Aga Khan Foundation (Other); Guttmacher Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2.4.8
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum hemorrhage; prevention; misoprostol; Uniject; oxytocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Experimental): 600 mcg oral misoprostol administered during the third stage of labor
  Interventions: Drug: misprostol
- UnijectTM (Experimental): 10 IU oxytocin delivered IM with UnijectTM during he third stage of labor
  Interventions: Device: UnijectTM

INTERVENTIONS:
Drug: misprostol — 600 mcg misoprostol oral
  Other Names: Cytotec
  Arms: Misoprostol
Device: UnijectTM — 10 IU oxytocin delivered intramuscularly with UnijectTM
  Arms: UnijectTM

SUMMARY:
This is a large, community-based, cluster-randomized trial to compare routine prophylactic use of 600 mcg oral misoprostol and 10 IU oxytocin delivered by UnijectTM intramuscularly during the third stage of labor.

DETAILED DESCRIPTION:
This study will assess the programmatic implications (including feasibility, acceptability, costs, risks and benefits) at the community level of the introduction of misoprostol and/or oxytocin in UnijectTM for the prevention of PPH and will help to identify the appropriate niche for both drugs.

ELIGIBILITY:
Inclusion Criteria:

* women delivering at home with a trained study provider who are able to provide informed consent

Exclusion Criteria:

* women with known contraindications to prostaglandins

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Mean change in hemoglobin | during 3rd trimester and 1-3 days postpartum
  To establish the comparable effectiveness of two technologies, individual pre- and post-delivery Hb measures will be taken to calculate change in Hb. This will be done using a Hemocue Hemoglobin machine + cuvette (HemoCue, Angelholm, Sweden). The Hemocue is a simple means of collecting Hb measures at the community-level where traditional laboratory techniques are not feasible.

SECONDARY OUTCOMES:
occurrence and management of side effects | 1 hour postpartum
  nausea, vomiting, diarrhea, shivering, fever
correct timing of drug administration | collected immediately following birth, verified 1-3 days postpartum
  administration of the drug after the birth of the baby and verifying no twin, before the expulsion of the placenta
change in hemoglobin ≥ 2 g/dL | during third trimester and 1-3 days postpartum
additional interventions | during birth and 1-3 days postpartum
  use of additional uterotonics, manual removal of placental fragments, etc
referrals | 1-3 days postpartum
  referral requested, transfers carried out, reasons for incomplete referrals/transfers
acceptability | 1-3 days postpartum
  acceptability according to woman of study medication, care received, side effects experienced

CONTACTS AND LOCATIONS:
Overall Officials: Ayisha R Diop, MPH, Principal Investigator — Gynuity Health Projects; Laura J Frye, MPH, Principal Investigator — Gynuity Health Projects; Yacouba Kone, M.D, Principal Investigator — The Aga Khan Foundation
Locations (1):
- Villages in Mopti, Mopti, Mali